CLINICAL TRIAL: NCT04460079
Title: Safety and Effectiveness Assessment of PeGagen® (Pegfilgrastim) in the Prevention of Chemotherapy-induced Febrile Neutropenia in Iranian Cancer Patients
Brief Title: Safety and Effectiveness Assessment of PeGagen® (Pegfilgrastim) in the Prevention of Chemotherapy-induced FN
Status: Completed | Type: Observational
Sponsor: Cinnagen (Industry)
Responsible Party: Sponsor
Other Study IDs: PEGAGEN.CIN.AJ.95 (IV)
Record Dates: First submitted 2020-06-27; First posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-05

CONDITIONS: Chemotherapy-induced Neutropenia
Keywords: Febrile neutropenia; Pegfilgrastim; Post-marketing surveillance; Chemotherapy-induced neutropenia; myelosuppressive chemotherapy
MeSH Terms: conditions — Febrile Neutropenia | interventions — pegfilgrastim

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Peg-filgrastim — PegaGen® was injected as a single subcutaneous dose after completion of cytotoxic chemotherapy
  Other Names: PegaGen®

SUMMARY:
The present study was an observational, multicenter, non-interventional, single arm, open label, PMS study conducted in Iran.

The primary objective of this study was safety assessment, including the rate of AEs. The secondary objective was the effectiveness evaluation in the prevention of chemotherapy-induced FN.

DETAILED DESCRIPTION:
The present study was an observational, multicenter, non-interventional, single arm, open label, PMS study conducted in Iran.

Data was gathered in two booklets, each containing information on four cycles of chemotherapy, which was filled by the designated physician. The duration of PegaGen® treatment was at the physicians' discretion based on the patient's condition.

The primary objective of this study was safety assessment, including the rate of AEs. The secondary objective was the effectiveness evaluation in the prevention of chemotherapy-induced FN.

This study was single arm and 654 subjects participated across various tumor types and regimens.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years,
* with the diagnosis of various types of cancers (such as lymphoma, breast, lung, testicular, prostate, ovary and gastrointestinal cancers), receiving first-line chemotherapy regimens with a high FN risk, which PegaGen® is injected due to physician decision.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving various tumor types and regimens with chemotherapy regimens of high FN risk, will be included.
Sampling Method: Non-Probability Sample
Enrollment: 654 (Actual)
Dates: Start 2016-03-29 (Actual); Primary Completion 2019-09-07 (Actual); Study Completion 2019-09-07 (Actual)

PRIMARY OUTCOMES:
Safety assessment, using incidence according to SOC and PT of AEs and SAEs | This outcome was assessed throughout the study, up to 8 chemotherapy cycles. The duration of treatment was at the physicians' discretion based on the patient's condition.
  Safety evaluation was reported using summary statistics. For each AE, data was summarized using incidence according to system organ class and preferred term of AEs and SAEs. Moreover, causality assessment was done and its results was reported by frequency and percentage.

SECONDARY OUTCOMES:
Effectiveness assessment: The frequency of neutropenia and neutropenic fever | This outcome was assessed throughout the study, up to 8 chemotherapy cycles. The duration of treatment was at the physicians' discretion based on the patient's condition.
  The frequency of neutropenia and neutropenic fever was reported

CONTACTS AND LOCATIONS:
Overall Officials: Arash Jenabian, Professor, Principal Investigator — Oncology & Hematology Dep., Booali Hosp., Islamic Azad University, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jenabian A, Ehsanpour A, Mortazavizadeh SMR, Raafat J, Razavi M, Khosravi A, Seifi S, Salimi B, Anjidani N, Kafi H. Evaluating the safety and effectiveness of PegaGen(R) (pegfilgrastim) for the prevention of chemotherapy-induced febrile neutropenia: a post-marketing surveillance study. Support Care Cancer. 2022 Oct;30(10):8151-8158. doi: 10.1007/s00520-022-07265-2. Epub 2022 Jul 6. PMID 35792924